CLINICAL TRIAL: NCT00723164
Title: Low Dose Fentanyl/Midazolam Improves Sevoflurane Induction in Adults
Brief Title: Premedication on Sevoflurane Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Sandra Lesage (resident), University of Montreal/Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05041
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Anesthesia
Keywords: Sevoflurane induction; Premedication; laryngeal mask airway; Anesthesia, inhalation [E03.155.197.197]
MeSH Terms: interventions — Fentanyl; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FM (Active Comparator): Premedication consisting of fentanyl 0.6 ug/kg and midazolam 9 ug/kg (FM), five minutes before tidal volume sevoflurane 8% induction with 6 L/min O2.
  Interventions: Drug: Fentanyl and Midazolam
- NaCl (Placebo Comparator): A 2.5 ml NaCL placebo (NaCl) IV, five minutes before tidal volume sevoflurane 8% induction with 6 L/min O2.
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Fentanyl and Midazolam — A combination of fentanyl 0.6 ug/kg and midazolam 9 ug/kg, to which NaCl was added to obtain a volume of 2.5 mL (group FM) injected IV, 5 minutes prior inhalation induction of anesthesia with sevoflurane
  Arms: FM
Drug: NaCl — NaCl 0.9% 2.5 ml intravenous (IV), 5 minutes prior inhalation induction of anesthesia with sevoflurane.
  Arms: NaCl

SUMMARY:
The goal of this study was to investigate the effects of fentanyl-midazolam premedication during sevoflurane induction pertaining to time to loss of eyelash reflex (LER), time and conditions of insertion of proseal laryngeal mask airway (PLMA), as well as cardio-respiratory data. Participants' anxiety level was also evaluated.

DETAILED DESCRIPTION:
Eighty adult patients undergoing minor surgery were randomized in a double-blind fashion. Each group received either a NaCL placebo (NaCl), or a premedication consisting of fentanyl 0,6 ug/kg and midazolam 9 ug/kg (FM), five minutes before tidal volume sevoflurane 8% induction with 6 L/min O2. Times to LER and LMA insertion were recorded. Adverse events were also noted. Systolic blood pressure (sBP), heart rate (HR), respiratory rate (RR) and tidal volume (Vt) were recorded at one-minute intervals. End-tidal sevoflurane (EtSevo) and end-tidal CO2 (EtCO2) were noted immediately following LMA insertion. Anxiety levels (0-10 verbal scale) were registered before and after premedication. Patients were contacted 24 hours postoperatively and were asked if they remembered the mask being applied to their face.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Minor elective surgery
* General anesthesia

Exclusion Criteria:

* Gastroesophageal reflux
* Exhibited a body mass index > 32 kg/m2
* Took sedative or opioid drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Impact of administering a combination of low doses of IV fentanyl and midazolam on time to loss of consciousness, and time of insertion of a laryngeal mask airway during sevoflurane induction. | 5 minutes after the premedication, each 30 seconds until the insertion of laryngeal mask airway

SECONDARY OUTCOMES:
Participants' cardiorespiratory status | 5 minutes after the premedication, at each minutes for 10 minutes
Patients' anxiety level | Before and after premedication and 24 hrs post op
Adverses events | 5 minutes after the premedication until the end of laryngeal mask insertion
Satisfaction | 24 hrs post op

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Drolet, MD, FRCPC, Study Director — Maisonneuve-Rosemont Hospital; Sandra Lesage, MD, Principal Investigator — Université de Montréal
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

REFERENCES:
- [Result] Joo HS, Perks WJ. Sevoflurane versus propofol for anesthetic induction: a meta-analysis. Anesth Analg. 2000 Jul;91(1):213-9. doi: 10.1097/00000539-200007000-00040. PMID 10866915
- [Result] Siddik-Sayyid SM, Aouad MT, Taha SK, Daaboul DG, Deeb PG, Massouh FM, Muallem MA, Baraka AS. A comparison of sevoflurane-propofol versus sevoflurane or propofol for laryngeal mask airway insertion in adults. Anesth Analg. 2005 Apr;100(4):1204-1209. doi: 10.1213/01.ANE.0000148166.29749.3B. PMID 15781547
- [Result] Ganatra SB, D'Mello J, Butani M, Jhamnani P. Conditions for insertion of the laryngeal mask airway: comparisons between sevoflurane and propofol using fentanyl as a co-induction agent. A pilot study. Eur J Anaesthesiol. 2002 May;19(5):371-5. doi: 10.1017/s0265021502000601. PMID 12095019
- [Result] Ti LK, Chow MY, Lee TL. Comparison of sevoflurane with propofol for laryngeal mask airway insertion in adults. Anesth Analg. 1999 Apr;88(4):908-12. doi: 10.1097/00000539-199904000-00041. PMID 10195546
- [Result] Hattori J, Yamakage M, Iwasaki S, Chen X, Tsujiguchi N, Namiki A. Usefulness of midazolam premedication for volatile induction of anesthesia in adults. J Anesth. 2001;15(2):117-9. doi: 10.1007/s005400170041. No abstract available. PMID 14566537
- [Result] Nishiyama T, Matsukawa T, Yokoyama T, Hanaoka K. Rapid inhalation induction with 7% sevoflurane combined with intravenous midazolam. J Clin Anesth. 2002 Jun;14(4):290-5. doi: 10.1016/s0952-8180(02)00361-6. PMID 12088814
- [Result] Sivalingam P, Kandasamy R, Madhavan G, Dhakshinamoorthi P. Conditions for laryngeal mask insertion. A comparison of propofol versus sevoflurane with or without alfentanil. Anaesthesia. 1999 Mar;54(3):271-6. doi: 10.1046/j.1365-2044.1999.00663.x. PMID 10364865
- [Result] Nathan N, Vandroux D, Benrhaiem M, Marquet P, Preux PM, Feiss P. Low alfentanil target-concentrations improve hemodynamic and intubating conditions during induction with sevoflurane. Can J Anaesth. 2004 Apr;51(4):382-7. doi: 10.1007/BF03018244. PMID 15064269
- [Result] Meaudre E, Boret H, Suppini A, Sallaberry M, Benefice S, Palmier B. Sufentanil supplementation of sevoflurane during induction of anaesthesia: a randomized study. Eur J Anaesthesiol. 2004 Oct;21(10):793-6. doi: 10.1017/s0265021504000079. PMID 15678734
- [Result] Muzi M, Colinco MD, Robinson BJ, Ebert TJ. The effects of premedication on inhaled induction of anesthesia with sevoflurane. Anesth Analg. 1997 Nov;85(5):1143-8. doi: 10.1097/00000539-199711000-00034. PMID 9356116
- [Result] Katoh T, Nakajima Y, Moriwaki G, Kobayashi S, Suzuki A, Iwamoto T, Bito H, Ikeda K. Sevoflurane requirements for tracheal intubation with and without fentanyl. Br J Anaesth. 1999 Apr;82(4):561-5. doi: 10.1093/bja/82.4.561. PMID 10472223
- [Result] Inagaki Y, Sumikawa K, Yoshiya I. Anesthetic interaction between midazolam and halothane in humans. Anesth Analg. 1993 Mar;76(3):613-7. doi: 10.1213/00000539-199303000-00029. PMID 8452276
- [Result] Ben-Shlomo I, abd-el-Khalim H, Ezry J, Zohar S, Tverskoy M. Midazolam acts synergistically with fentanyl for induction of anaesthesia. Br J Anaesth. 1990 Jan;64(1):45-7. doi: 10.1093/bja/64.1.45. PMID 2302375
- [Result] Plastow SE, Hall JE, Pugh SC. Fentanyl supplementation of sevoflurane induction of anaesthesia. Anaesthesia. 2000 May;55(5):475-8. doi: 10.1046/j.1365-2044.2000.01268.x. PMID 10792142
- [Result] Hall JE, Stewart JI, Harmer M. Single-breath inhalation induction of sevoflurane anaesthesia with and without nitrous oxide: a feasibility study in adults and comparison with an intravenous bolus of propofol. Anaesthesia. 1997 May;52(5):410-5. doi: 10.1111/j.1365-2044.1997.091-az0086.x. PMID 9165957
- [Result] Siau C, Liu EH. Nitrous oxide does not improve sevoflurane induction of anesthesia in adults. J Clin Anesth. 2002 May;14(3):218-22. doi: 10.1016/s0952-8180(02)00349-5. PMID 12031757
- [Result] Philip BK, Lombard LL, Roaf ER, Drager LR, Calalang I, Philip JH. Comparison of vital capacity induction with sevoflurane to intravenous induction with propofol for adult ambulatory anesthesia. Anesth Analg. 1999 Sep;89(3):623-7. doi: 10.1097/00000539-199909000-00014. PMID 10475291
- [Result] Yogendran S, Prabhu A, Hendy A, McGuire G, Imarengiaye C, Wong J, Chung F. Vital capacity and patient controlled sevoflurane inhalation result in similar induction characteristics. Can J Anaesth. 2005 Jan;52(1):45-9. doi: 10.1007/BF03018579. PMID 15625255
- [Result] Baker CE, Smith I. Sevoflurane: a comparison between vital capacity and tidal breathing techniques for the induction of anaesthesia and laryngeal mask airway placement. Anaesthesia. 1999 Sep;54(9):841-4. doi: 10.1046/j.1365-2044.1999.00949.x. PMID 10460554
- [Result] Nathan N, Bazin JE, Cros AM. [Inhalation induction]. Ann Fr Anesth Reanim. 2004 Sep;23(9):884-99. doi: 10.1016/j.annfar.2004.07.017. French. PMID 15471636
- [Result] Kelly RE, Hartman GS, Embree PB, Sharp G, Artusio JF Jr. Inhaled induction and emergence from desflurane anesthesia in the ambulatory surgical patient: the effect of premedication. Anesth Analg. 1993 Sep;77(3):540-3. doi: 10.1213/00000539-199309000-00019. PMID 8368553
- [Result] Pancaro C, Giovannoni S, Toscano A, Peduto VA. Apnea during induction of anesthesia with sevoflurane is related to its mode of administration. Can J Anaesth. 2005 Jun-Jul;52(6):591-4. doi: 10.1007/BF03015767. PMID 15983143
- [Result] Joo HS, Perks WJ, Belo SE. Sevoflurane with remifentanil allows rapid tracheal intubation without neuromuscular blocking agents. Can J Anaesth. 2001 Jul-Aug;48(7):646-50. doi: 10.1007/BF03016197. PMID 11495870
- [Result] Cardinal V, Martin R, Tetrault JP, Colas MJ, Gagnon L, Claprood Y. [Severe bradycardia and asystole with low dose sufentanil during induction with sevoflurane: a report of three cases]. Can J Anaesth. 2004 Oct;51(8):806-9. doi: 10.1007/BF03018453. French. PMID 15470169
- [Result] Wang J, Winship S, Russell G. Induction of anaesthesia with sevoflurane and low-dose remifentanil: asystole following laryngoscopy. Br J Anaesth. 1998 Dec;81(6):994-5. doi: 10.1093/bja/81.6.994-a. No abstract available. PMID 10211042
- [Result] Kurdi O, Deleuze A, Marret E, Bonnet F. Asystole during anaesthetic induction with remifentanil and sevoflurane. Br J Anaesth. 2001 Dec;87(6):943. No abstract available. PMID 11878707
- [Result] Le May S, Hardy JF, Taillefer MC, Dupuis G. Measurement of patient satisfaction. Anesth Analg. 1999 Jul;89(1):255. doi: 10.1097/00000539-199907000-00047. No abstract available. PMID 10389815
- [Derived] Lesage S, Drolet P, Donati F, Racine S, Fortier LP, Audy D. Low-dose fentanyl-midazolam combination improves sevoflurane induction in adults. Can J Anaesth. 2009 Oct;56(10):733-9. doi: 10.1007/s12630-009-9150-6. Epub 2009 Jul 30. PMID 19641980